CLINICAL TRIAL: NCT06941077
Title: Relative Bioavailability of New Formulations of INCB057643 Tablets Administered Orally in Healthy Participants
Brief Title: A Study to Evaluate the Relative Bioavailability of New Formulations of INCB057643 Tablets Administered Orally in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: INCB057643-111
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers
Keywords: INCB057643
MeSH Terms: interventions — INCB057643

STUDY DESIGN:
Intervention Model Description: Cohorts 1-3 are single dose, and Cohort 4 is single dose, 2-way crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cohort 1: Dose Treatment A (Experimental): INCB057643 will be administered at protocol defined dose.
  Interventions: Drug: INCB057643
- Cohort 2: Dose Treatment B (Experimental): INCB057643 will be administered at protocol defined dose.
  Interventions: Drug: INCB057643
- Cohort 3: Dose Treatment C (Experimental): INCB057643 will be administered at protocol defined dose.
  Interventions: Drug: INCB057643
- Cohort 4: Dose Treatment D (Experimental): INCB057643 will be administered at protocol defined dose.
  Interventions: Drug: INCB057643
- Cohort 4: Dose Treatment E (Experimental): INCB057643 will be administered at protocol defined dose.
  Interventions: Drug: INCB057643

INTERVENTIONS:
Drug: INCB057643 — Tablet

SUMMARY:
The purpose of this study is to evaluate the Relative Bioavailability of New Formulations of INCB057643 Tablets Administered Orally in Healthy Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Aged 18 to 55 years, inclusive, at the time of signing the ICF.
* BMI within the range of 18.0 to 30.0 kg/m2 inclusive. Note: Up to 25% of the participants in each cohort may be enrolled with a BMI > 30 to ≤ 32.0 kg/m2.
* No clinically significant findings on screening evaluations (clinical, laboratory, and ECG).
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of uncontrolled or unstable respiratory, renal, GI, endocrine, hematopoietic, psychiatric, and/or neurological disease within 6 months of screening.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension.
* High blood pressure (systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* History or presence of an abnormal ECG before screening and check-in that, in the investigator's opinion, is clinically significant, such as a QTcF interval > 450 milliseconds, QRS interval > 120 milliseconds, or PR interval > 220 milliseconds.
* History or presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn disease or chronic pancreatitis).
* Hepatic transaminases (ALT and AST), ALP, or total bilirubin > 1.25 × the laboratory-defined ULN at screening and check-in, confirmed by repeat testing (except participants with Gilbert disease, for which total bilirubin must be ≤ 2.0 × ULN).
* Any major surgery within 4 weeks of screening.
* Current or recent (within 3 months of screening) clinically significant GI disease or surgery (including cholecystectomy and excluding appendectomy) that could affect the absorption of study drug.
* Donation of blood to a blood bank or participation in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for donation of plasma only).
* Positive test for HBV, HCV, or HIV. Participants whose results are compatible with prior immunization for or immunity due to infection with HBV may be included at the discretion of the investigator.
* History of significant alcohol use, defined as regular alcohol consumption > 21 units per week for males and > 14 units for females (1 unit = 8 ounces of beer or a 25-mL shot of 40% spirit, 1.5 to 2 units = 125-mL glass of wine, depending on type).
* Positive urine or breath test for ethanol or positive urine or serum screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug or investigational product study.
* History of tobacco or nicotine-containing product use within 1 month of screening.
* Use of prescription drugs (including hormonal contraceptives) within 14 days of study drug administration or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations) within 7 days of study drug administration. However, occasional and standard-dose acetaminophen and ibuprofen and standard-dose vitamins are permitted. Megadose vitamins or supplements are not permissible.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2025-05-12 (Actual); Primary Completion 2025-06-03 (Actual); Study Completion 2025-06-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics Parameter (PK): Cmax of INCB057643 | Up to Day 10
  Defined as maximum observed plasma concentration of INCB057643.
Pharmacokinetics Parameter: AUC(0-last) of INCB057643 | Up to Day 10
  Defined as area under the single-dose serum concentration-time curve from time = 0 to the last measurable concentration at time of INCB057643.
Pharmacokinetics Parameter: AUC 0-∞ of INCB057643 | Up to Day 10
  Defined as the area under the single-dose serum concentration-time curve extrapolated to time of infinity of INCB057643.

SECONDARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Events (TEAEs) | Up to Day 26
  Defined as adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug.
Pharmacokinetics Parameter: Tmax of INCB057643 | Up to Day 10
  Defined as the time to reach the maximum plasma concentration of INCB057643.
Pharmacokinetics Parameter: t1/2 of INCB057643 | Up to Day 10
  Defined as the apparent terminal phase disposition half-life of INCB057643.
Pharmacokinetics Parameter: CL/F INCB057643 | Up to Day 10
  Defined as the apparent oral dose clearance of INCB057643.
Pharmacokinetics Parameter: V2/F of INCB057643 | Up to Day 10
  Defined as the apparent oral dose volume of distribution of INCB057643.
Pharmacokinetics Parameter: λz of INCB057643 | Up to Day 10
  Defined as apparent terminal-phase disposition rate constant of INCB057643.
Pharmacokinetics Parameter: %AUCexp of INCB057643 | Up to Day 10
  Defined as percentage of AUC0-∞ due to extrapolation from the time of last quantifiable concentration to infinity of INCB057643.

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Study Monitor, Study Director — Incyte Corporation
Locations (1):
- Celerion, Inc, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Study to Evaluate the Relative Bioavailability of New Formulations of INCB057643 Tablets Administered Orally in Healthy Participants — https://www.incyteclinicaltrials.com/trials/INCB057643-111